CLINICAL TRIAL: NCT06035471
Title: Can we Use a Simple Blood Test to Reduce Unnecessary Adverse Effects From Radiotherapy by Timely Identification of Radiotherapy-resistant Rectal Cancers? MeD-Seq Rectal Study
Status: Not yet recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, C. Verhoef, Professor, Erasmus Medical Center
Other Study IDs: Med-Seq Rectal
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Pathological Response Rate, Circulating Tumour DNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MeD-seq — MeD-seq analyse: DNA treatment bisulfite --> unmethylated C-nucleotide trabsformed in uracil.--> PCR --> next generation sequencing (NGS) --> localization methylated nucleotides (enzym LpnPI).

SUMMARY:
Chemoradiation therapy (CRT) followed by surgery is currently the standard of care to treat patients with locally advanced rectal cancer (LARC). CRT reduces local recurrences, but is associated with significant damage to the surrounding healthy tissue that can severely impact quality of life. Additionally, a proportion of patients (hardly) benefit from CRT. We aim to develop a diagnostic innovation, which can enable a more selective and thereby more effective use of the available therapies for rectal cancer patients.

The objective of this study is to investigate whether patients can be identified who will response to CRT prior to start of the CRT in rectal cancer and therefore avoid possible severe side effects in patients who will not reponse on CRT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically confirmed rectal adenocarcinoma
* Scheduled for neoadjuvant chemoradiation
* Written informed consent.

Exclusion Criteria:

* Scheduled to another neoadjuvant schedule that comprises systemic chemotherapy or short-course radiation
* Not able to read or understand Dutch language or mentally not capable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally advanced rectal cancer patients scheduled for preoperative chemoradiation
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
cfDNA methylation markers | 4 years

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mens DM, van Rees JM, Wilting SM, Verhoef C. Can we use a simple blood test to reduce unnecessary adverse effects from radiotherapy by timely identification of radiotherapy-resistant rectal cancers? MeD-Seq rectal study protocol. BMC Cancer. 2023 Dec 4;23(1):1187. doi: 10.1186/s12885-023-11671-y. PMID 38049783